CLINICAL TRIAL: NCT06176040
Title: A Pilot Phase 2A Study to Examine the Preliminary Efficacy, Safety and PK of TAVO101 in Patients with Moderate to Severe Atopic Dermatitis (AD)
Brief Title: A Study of TAVO101 in Atopic Dermatitis Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tavotek Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 59870004
Record Dates: First submitted 2023-12-10; First posted 2023-12-19 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Eczema; TAVO101
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TAVO101: High Dose (Experimental): TAVO101 IV Infusion given as loading dose, every 2 months (Q2M), every 3 months (Q3M).
  Interventions: Drug: TAVO101
- TAVO101: Medium Dose (Experimental): TAVO101 IV Infusion given as loading dose and Q3M.
  Interventions: Drug: TAVO101
- TAVO101: Medium Low Dose (Experimental): TAVO101 IV Infusion given as loading dose and Q2M.
  Interventions: Drug: TAVO101
- TAVO101: Low Dose Control (Experimental): TAVO101 IV Infusion given as loading dose and Q2M.
  Interventions: Drug: TAVO101

INTERVENTIONS:
Drug: TAVO101 — TAVO101 IV Infusion.

SUMMARY:
This is a Phase 2 pilot study to examine the preliminary efficacy, safety and PK of TAVO101 in adult patients with moderate and severe AD.

DETAILED DESCRIPTION:
This is a Phase 2 pilot study to examine the preliminary efficacy, safety and PK of TAVO101 in adult patients with moderate and severe AD.

The total treatment and observation period is 24 weeks in duration of which the last dose of drug will be given by Week 16, leaving the last 8 weeks as an extra period for safety monitoring. Approximately 20 patients will be randomized in a 1:1:1:1 ratio to receive intravenous treatment of TAVO101 in 4 different dosing schemes. TAVO101 in 210-420 mg flat dose administered every 4 to 12 weeks will be tested to examine the preliminary effect of different dose and dosing interval in managing atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 75 years old
2. Body weight range of ≥ 50 kg and ≤ 110 kg, inclusive, and a body mass index (BMI) ≥ 18.0 and ≤ 31.0 kg/m2
3. A diagnosis of chronic AD and has been present for at least 6 months before the screening visit.
4. AD Diagnosis confirmed by the Eichenfield revised criteria of Hannifin and Rajka at the screening visit.
5. All the following conditions must be met to fit the Severe AD classification:

   * ≥10% body surface area (BSA) of AD involvement at the screening and baseline visits.
   * Eczema Area and Severity Index (EASI) score ≥ 11 to be considered moderate AD and ≥16 to be considered severe AD at the screening and baseline visits.
   * Investigator's Global Assessment (IGA) score ≥3 at the screening and baseline visits.
   * Serum IgE concentration ≥150 kU/L at the screening visit.
   * History of intolerant or inadequate response to a stable (1 month) regimen of topical corticosteroids or calcineurin inhibitors as treatment for AD within 12 months before the screening visit.
6. Subjects must have applied a stable dose of emollient twice daily (or more, as needed) for at least 7 days before randomization.
7. No clinically significant abnormality on the basis of medical/medication history or physical examination.
8. Willing and able to comply with clinic visits and study-related procedures.
9. Patient able to read and understand, and willing to sign the informed consent form (ICF).
10. Females of childbearing potential who are sexually active with a non-sterilized male partner must use highly effective contraception from enrollment and must agree to continue using such precautions through to study end. Females of childbearing potential are defined as those who are not surgically sterile or post-menopausal. A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly.
11. Males who are sexually active and whose partners are females of childbearing potential must agree to use condoms (unless surgically sterile) from Screening through 60 days after the last dose of study drug, and their partners must be willing to use a highly effective method of contraception from Screening through 60 days after the last dose of study drug.

Exclusion Criteria:

1. Active dermatologic conditions, which may confound the AD diagnosis or treatment assessment.
2. Known active allergic or irritant contact dermatitis.
3. Systemic treatment for AD with an immunosuppressive / immunomodulating substance within 4 weeks prior to the baseline visit, e.g., azathioprine, methotrexate, cyclosporine, mycophenolate-mofetil, tacrolimus, interferon-γ, or phototherapy (narrow band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + ultraviolet A [PUVA]).)
4. Treatment with topical phosphodiesterase-4 (PDE-4) inhibitor, topical corticosteroids (TCS), topical calcineurin inhibitors (TCI), and other topical AD treatments within 2 weeks before the baseline visit.
5. Treatment of AD with a medical device (eg, Atopiclair®, MimyX®, Epicerum®, Cerave®, etc) within 1 week before the baseline visit.
6. Treatment with allergen immunotherapy within 6 months before the baseline visit.
7. Patients with severe respiratory or autoimmune diseases that require chronic systemic corticosteroid or immuno-suppressive therapies for disease management.
8. Chronic or acute infection requiring treatment with oral or IV antibiotics, anti-virals, anti-parasitics, anti-protozoals, or anti-fungals within 4 weeks before the screening visit or superficial skin infections within 1 week before the screening visit.
9. Treatment with any marketed or investigational biologic agent within 3 months or 5 half-lives prior to baseline, whichever is longer; Or receipt of any investigational non-biologic agent within 3 months or 5 half-lives prior to baseline, whichever is longer.
10. Patients who have received a live or attenuated vaccine within 8 weeks prior to baseline. Receipt of inactive/killed vaccinations (eg, inactive influenza) is allowed provided they are not administered within 1 week before/after any study visit.
11. Positive hepatitis B surface antigen or hepatitis C virus antibody serology. Patients with a history of hepatitis B vaccination without history of hepatitis B are allowed to enroll.
12. A positive human immunodeficiency (HIV) virus test at screening or patient taking antiretroviral medications.
13. Diagnosis of a helminth parasitic infection within 6 months prior to screening that has not been treated with, or has failed to respond to standard of care therapy.
14. Patients who, in the opinion of the investigator, have a positive Quanti FERON tuberculosis Gold (QFT-G) test for tuberculosis (TB) during screening or have evidence of active treated or untreated TB. Patients with an indeterminate QFT-G result may be enrolled if they have all of the following: a). No symptoms of TB; b) No known exposure to a case of active TB; c) No evidence of active TB on chest radiograph within 3 months prior to baseline. Patients with an indeterminate QFT-G result will have repeat QFT-G testing at Week 12.
15. History of cancer, except for basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success ≥12 months prior to screening or other malignancies treated with apparent success ≥5 years prior to screening.
16. History of anaphylaxis or severe infusion related reaction (IRR) following any biologic therapy.
17. Any clinically relevant abnormal findings in physical electrocardiogram examination, vital signs, hematology, clinical chemistry, or urinalysis during screening, which in the opinion of the investigator may compromise the patient's safety, interfere with evaluation of the study treatment or reduce the patient's ability to participate in the study. Evidence of active liver disease, including jaundice or aspartate transaminase, alanine transaminase, or alkaline phosphatase greater than twice the upper limit of normal.
18. Major surgery within 8 weeks prior to screening or planned in-patient surgery or hospitalization during the study period.
19. Use of a tanning booth/parlor within 8 weeks before the screening visit.
20. Pregnant or breast-feeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who achieve a 50% Reduction From Baseline in Eczema Area and Severity (EASI 50) at Week 16 | Baseline to Week 16
  The EASI evaluates 4 natural anatomical regions for severity and extent of key disease signs and focuses on key acute and chronic signs of inflammation (ie, erythema, induration/papulation, excoriation, and lichenification).

SECONDARY OUTCOMES:
Proportion of Patients With Investigator's Global Assessment (IGA) Score of 0 (Clear) or 1 (Almost Clear) at Week 16 | Baseline to Week 16
  The IGA allows investigators to assess overall disease severity at 1 given time point and consists of a 6-point severity scale from clear to severe disease
  0 = clear
  1. = almost clear
  2. = mild disease
  3. = moderate disease
  4. = severe disease
  5. = very severe disease
Proportion of patients who achieve a 75% Reduction From Baseline in Eczema Area and Severity (EASI 75) at Week 16 | Baseline to Week 16
  The EASI evaluates 4 natural anatomical regions for severity and extent of key disease signs and focuses on key acute and chronic signs of inflammation (ie, erythema, induration/papulation, excoriation, and lichenification).
Change from Baseline in Scoring Atopic Dermatitis (SCORAD) at Week 16 | Baseline to Week 16
  The SCORAD is a clinical tool for assessing the severity (ie, extent, intensity) of atopic dermatitis (AD). The tool evaluates the extent and intensity of the AD lesions, along with subjective symptoms (Kunz et al, 1997). The total score ranges from 0 to 103, with higher values indicating more severe disease. A negative change from baseline indicates an improvement in severity of disease.
Change from Baseline of Pruritus Numerical Rating Scale (NRS) at Week 16 | Baseline to Week 16
  The Peak Pruritus NRS is a single-item scale used by patients to rate itch severity in moderate-to-severe atopic dermatitis. It ranges from 0 (no itch) to 10 (worst imaginable itch), with a significant response defined as a 2-4 point change.
Incidence of Treatment Emergent Adverse Events (TEAES) from Baseline to Week 24 | Baseline to Week 24
  To investigate the safety and tolerability of TAVO101 in AD patients.
Cmax (Maximum observed serum concentration) of TAVO101 | Baseline to Week 24
  To investigate the pharmacokinetics (PK) in TAVO101.
Immunogenicity of TAVO101 | Baseline to Week 24
  To investigate the incidence of anti-drug antibodies (ADA) following dosing of TAVO101.

CONTACTS AND LOCATIONS:
Overall Officials: Penelope Montgomery, MD, Principal Investigator — Optimal Clinical Trials
Locations (2):
- Royal Melbourne Hospital, Parkville, Victoria, Australia
- Optimal Clinical Trials, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No